CLINICAL TRIAL: NCT04835740
Title: Effects of High-intensity Interval Aerobic Training on Balance, Walking Capacity, and Quality of Life in Patients With Sub-acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akhtar Saeed Medical and Dental College (Other)
Responsible Party: Principal Investigator, Memoona Azhar, Physiotherapist, Akhtar Saeed Medical and Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/ASCRH/0006/2020
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Stroke, Ischemic; Cerebrovascular Accident
Keywords: Cerebrovascular accident; Treadmill Training; High-intensity interval training; Walking capacity.
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Rehabilitation (Active Comparator): Based on the functional capacity of each participant, customized Aerobic exercise plan was designed by the on-site physiotherapist.
  Interventions: Other: High intensity Interval Training
- Combined Training (conventional rehabilitation plus high-intensity interval training): (Experimental): The patients received 40 minutes of High intensity interval treadmill training in addition to their normal conventional rehabilitation.
  Interventions: Other: High intensity Interval Training

INTERVENTIONS:
Other: High intensity Interval Training — All the participants underwent 5 weeks of High intensity interval training.

SUMMARY:
Hemiplegia is one of the most common sequelae of stroke. Stroke is the leading cause of disability in adults all around the world. Stroke survivors can suffer several neurological impairments and deficits which have an important impact on patient's quality of life and which increase the costs for health and social services. After stroke, impairments in ADLs and functional status, deterioration in health related quality of life can be seen.

The purpose of this study is to Determine the effect of Aerobic exercise training on Balance, Walking capacity and quality of life in sub-acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age.
* Ischemic Stroke that occurred in the recent 3 months.
* Who can walk independently or by using assistive device.
* Have a minimum Chedoke McMaster Stroke Assessment (CMSA) leg impairment score of 3 but less than 7.

Exclusion Criteria:

* Patients were excluded from the study if they have a stroke that occurs more than 3 months.
* Hemorrhagic Stroke.
* If resting blood pressure more than 160/100 even after taking medications
* Have by-pass surgery in recent 3 months.
* Other musculoskeletal problems which restrict the patient's ability to do aerobic activity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
6 Minute walk Test | 5 weeks
  To determine the cardiorespiratory fitness of individual after sub-acute stroke.

SECONDARY OUTCOMES:
Berg Balance test and rating scale | 5 weeks
  The scale is used to determine the Balance and stability of patient. Total score of the scale is 56. A score of < 45 indicates individuals may be at greater risk of falling.
Stroke Impact scale | 5 weeks
  The scale is used to measure the impairment and quality of life after stroke. The scale consists of 8 domains. In this study, only 4 domains related to hand function ,strength, mobility and Activity of daily living were used.The maximum score is 140.

CONTACTS AND LOCATIONS:
Locations (1):
- Akhtar Saeed Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided